CLINICAL TRIAL: NCT00429936
Title: A Phase II Multicenter, Randomized, Double-Masked, Placebo-Controlled, Dose-Comparison Study of the Safety and Efficacy of Fenretinide in the Treatment of Geographic Atrophy in Subjects With Age-Related Macular Degeneration
Brief Title: Study of Fenretinide in the Treatment of Geographic Atrophy Associated With Dry Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sirion Therapeutics, Inc. (Industry)
Collaborators: ReVision Therapeutics, Inc. (Other)
Responsible Party: ReVision Therapeutics, Inc., ReVision Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRFR-001
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Geographic Atrophy; Dry Age Related Macular Degeneration
Keywords: Dry Age Related Macular Degeneration; Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — Fenretinide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 100 mg fenretinide softgel capsules (Active Comparator): Three (3) 100-mg fenretinide softgel capsules
  Interventions: Drug: Fenretinide
- Fenretinide and placebo softgel capsules (Active Comparator): One (1) 100-mg fenretinide softgel capsule and two (2) placebo softgel capsules
  Interventions: Drug: Fenretinide
- Placebo softgel capsules (Placebo Comparator): Three (3) placebo softgel capsules
  Interventions: Drug: Fenretinide

INTERVENTIONS:
Drug: Fenretinide — Once daily 30 minutes after the evening meal for 24 months

SUMMARY:
The purpose of this phase II study is to determine the efficacy of fenretinide in the treatment of geographic atrophy (GA) in subjects with the dry form of age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* males or females, 50 to 89 years of age
* must have GA from AMD in one or both eyes

Exclusion Criteria:

* GA due to any disease other than AMD (eg, drug-induced)

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2006-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
GA lesion progression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roger Vogel, MD, Study Director — ReVision Therapeutics Advisor

REFERENCES:
- [Derived] Yeong JL, Loveman E, Colquitt JL, Royle P, Waugh N, Lois N. Visual cycle modulators versus placebo or observation for the prevention and treatment of geographic atrophy due to age-related macular degeneration. Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD013154. doi: 10.1002/14651858.CD013154.pub2. PMID 33331670